CLINICAL TRIAL: NCT06061237
Title: Effects of Aerobic Thai Dance on Gait, Balance and Sudomotor Function in Patient With Diabetic Peripheral Neuropathy
Brief Title: Effects of Aerobic Thai Dance in Patient With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Thammarat Koksungnoen, Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0151/65
Record Dates: First submitted 2023-08-27; First posted 2023-09-29 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Exercise Addiction; Diabetic Neuropathies
Keywords: Diabetes Mellitus; Diabetic Peripheral Neuropathy; Thai Dance; Gait; Balance; Sudomotor Function; DPN; Exercise
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Thai dance exercise intervention (Experimental): Aerobic Thai dance exercise 60 minute per times, 3 times per weeks of 12 weeks.
  Interventions: Other: Aerobic Thai dance exercise
- Control (No Intervention): Give advice on exercise.

INTERVENTIONS:
Other: Aerobic Thai dance exercise — Aerobic Thai dance exercise 60 minute per times, 3 times per weeks of 12 weeks. Aerobic exercise of modulate intensity (12-13 Borg's RPE)
  Arms: Aerobic Thai dance exercise intervention

SUMMARY:
The goal of this type of study is clinical trial. This to learn about effects of applied aerobic Thai dance exercise on gait balance and sudomotor function in patient with diabetic peripheral neuropathy. Test variables of gait, balance, function of sudomotor, Physiological data such as pulse, blood pressure, body composition, ankle and leg muscle strength, compare with control and experimental group in diabetes with peripheral neuropathy.

The main question Question 1: Dose Applied aerobic Thai dance exercise affects gait and balance in diabetic patients with peripheral neuropathy? Question 2: Does applied aerobic Thai dance exercise affect sudomotor function in diabetic patients with peripheral neuropathy? Participants will divided into 2 groups: the control group and the experimental group. By randomly sampling 22 people from each group

1. The control group was advised to exercise at home for a period of 12 weeks.
2. The experimental group participated in Applied aerobic Thai dance exercise 60 minutes per session, 3 times per week, for a period of 12 weeks.

After 12 weeks, variable data were collected and to compare within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes between the ages of 60 and 75.
* The BMI index is between 18.5 - 29.9 kg/m2.
* MNSI score between 2.5 - 7.5 points.
* There were no exercise-related complications from the PAR -Q assessment.
* Light to moderate level of physical activity.
* Not being a person with severe optic neuropathy (Severe-NPDR and Severe-PDR).
* No wounds or infections on the feet.
* No musculoskeletal abnormalities.
* Not being a Pacemaker Implantation Person, No History of Heart Failure, Evaluated New York Heart Association Classification (NYHA) not over Functional Class II, If CAD must be treated, No history of Atrial Fibrillation severely wrong.
* The doctor did not have a plan to adjust the medication in the last 3 months.

Exclusion Criteria:

* MNSI score greater than or equal to 8 points or more.
* Participants lacked more than 20 percent of their exercise program.
* Participants had foot ulcers and infections during the experiment.
* Vitamins B1, 6 and 12 were taken during the trial.
* The subject withdrew from the experiment.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Gait Speed | Baseline and 12 weeks
  Gait Speed will be measured by Strideway in centimeter per seconds (cm/sec).
Step length | Baseline and 12 weeks
  Step length will be measured by Strideway in centimeter (cm).
Single Support | Baseline and 12 weeks
  Single Support will be measured by Strideway in seconds (sec).
Double Support | Baseline and 12 weeks
  Double Support will be measured by Strideway in seconds (sec).
Cadence | Baseline and 12 weeks
  Cadence will be measured by Strideway in steps per minute (steps/minute).
Postural Stability Testing | Baseline and 12 weeks
  Postural Stability Testing will be measured by Biodex balance system in score.
Modified Clinical Test of Sensory Interaction in Balance (M-CTSIB) | Baseline and 12 weeks
  Modified Clinical Test of Sensory Interaction in Balance (M-CTSIB) will be measured by Biodex balance system in score.
Limits of Stability (LOS) | Baseline and 12 weeks
  Limits of Stability (LOS) will be measured by Biodex balance system in score.
Time up and go test | Baseline and 12 weeks
  Functional balance test will be measured by Time up and go test in seconds.
Functional reach test | Baseline and 12 weeks
  Functional balance test will be measured by Functional reach test in centimeter.

SECONDARY OUTCOMES:
Sudomotor function | Baseline and 12 weeks
  Sudomotor function testing feet and hands will be measured by Sudoscan in microsiemens (µS).
Leg muscle strength | Baseline and 12 weeks
  Leg muscle strength testing will be measured by Isokinetic dynamometer in newton meter (Nm).
Ankle muscle strength | Baseline and 12 weeks
  Ankle Muscle strength testing will be measured by Hand-held dynamometry in kilogram (Kg).
Michigan Neuropathy Screening Instrument (MNSI) | Baseline and 12 weeks
  Questionnaire variables will be measured by Michigan Neuropathy Screening Instrument (MNSI) in score. The scale's range in score is from 0 to 13. Cut off greater than or equal to 2 scores and a low score represents mild neuropathy, whereas a high score represents severe neuropathy.
Short-form McGill Pain Questionnaire (SF-MPQ) | Baseline and 12 weeks
  Questionnaire variables will be measured by Short-form McGill Pain Questionnaire (SF-MPQ) in score. The scale's range in score is from 0 to 60. A low score represents no pain, whereas a high score represents worse pain.
Neurological symptom score (NSS) | Baseline and 12 weeks
  Questionnaire variables will be measured by Neurological symptom score (NSS) in score. The scale's range in score is from 0 to 18. A low score represents mild neuropathic symptoms, whereas a high score represents severe neuropathic symptoms.
Foot Pain Manikin | Baseline and 12 weeks
  Questionnaire variables will be measured by Foot Pain Manikin in score. The scale's range in score is from 0 to 50. A low score represents no area of pain, whereas a high score represents a wide area of pain.
Falls Efficacy Scale International (FES-I) | Baseline and 12 weeks
  Questionnaire variables will be measured by Falls Efficacy Scale International (FES-I) in score. The scale's range in score is from 16 to 64. A low score represents no concern about falling, whereas a high score represents severe concern about falling.
Fasting Plasma Glucose (FPG) | Baseline and 12 weeks
  Fasting Plasma Glucose (FPG) will be measured by medical technician in faculty of Allied Health Sciences Chulalongkorn University in milligrams per deciliter (mg/dL).
Hemoglobin A1c (HbA1C) | Baseline and 12 weeks
  Hemoglobin A1c (HbA1C) will be measured by medical technician in faculty of Allied Health Sciences Chulalongkorn University in percentage.
High Density Lipoprotein (HDL) | Baseline and 12 weeks
  High Density Lipoprotein (HDL) will be measured by medical technician in faculty of Allied Health Sciences Chulalongkorn University in milligrams per deciliter (mg/dL).
Low Density Lipoprotein (LDL) | Baseline and 12 weeks
  Low Density Lipoprotein (LDL) will be measured by medical technician in faculty of Allied Health Sciences Chulalongkorn University in milligrams per deciliter (mg/dL).
Blood pressure | Baseline and 12 weeks
  Blood pressure will be measured by Sphygmomanometer in mmHg.
Resting heart rate | Baseline and 12 weeks
  Resting heart rate will be measured by Sphygmomanometer in Times per minute (Times/ minute).
Weight | Baseline and 12 weeks
  Weight will be measured by Body Composition Analyzer in kilogram (kg).
Height | Baseline and 12 weeks
  Height will be measured by Body Composition Analyzer in centimeter (cm).
Body mass index (BMI) | Baseline and 12 weeks
  Weight and height will be combined to report Body mass index (BMI) in kg/m^2.
Body fat | Baseline and 12 weeks
  Body fat index will be measured by Dexa Scan in percentage.
Muscle mass | Baseline and 12 weeks
  Muscle mass index will be measured by Dexa Scan in kilogram (kg).

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn university, Bangkok, Thailand

REFERENCES:
- [Background] Adler AI, Boyko EJ, Ahroni JH, Smith DG. Lower-extremity amputation in diabetes. The independent effects of peripheral vascular disease, sensory neuropathy, and foot ulcers. Diabetes Care. 1999 Jul;22(7):1029-35. doi: 10.2337/diacare.22.7.1029. PMID 10388962
- [Background] Ahn S, Song R. Effects of Tai Chi Exercise on glucose control, neuropathy scores, balance, and quality of life in patients with type 2 diabetes and neuropathy. J Altern Complement Med. 2012 Dec;18(12):1172-8. doi: 10.1089/acm.2011.0690. Epub 2012 Sep 17. PMID 22985218
- [Background] Akbari M, Jafari H, Moshashaee A, Forugh B. Do diabetic neuropathy patients benefit from balance training? J Rehabil Res Dev. 2012;49(2):333-8. doi: 10.1682/jrrd.2010.10.0197. PMID 22773533
- [Background] Alam U, Riley DR, Jugdey RS, Azmi S, Rajbhandari S, D'Aout K, Malik RA. Diabetic Neuropathy and Gait: A Review. Diabetes Ther. 2017 Dec;8(6):1253-1264. doi: 10.1007/s13300-017-0295-y. Epub 2017 Sep 1. PMID 28864841
- [Background] Albright A, Franz M, Hornsby G, Kriska A, Marrero D, Ullrich I, Verity LS. American College of Sports Medicine position stand. Exercise and type 2 diabetes. Med Sci Sports Exerc. 2000 Jul;32(7):1345-60. doi: 10.1097/00005768-200007000-00024. PMID 10912903
- [Background] Baker LB. Physiology of sweat gland function: The roles of sweating and sweat composition in human health. Temperature (Austin). 2019 Jul 17;6(3):211-259. doi: 10.1080/23328940.2019.1632145. eCollection 2019. PMID 31608304
- [Background] Billot M, Handrigan GA, Simoneau M, Corbeil P, Teasdale N. Short term alteration of balance control after a reduction of plantar mechanoreceptor sensation through cooling. Neurosci Lett. 2013 Feb 22;535:40-4. doi: 10.1016/j.neulet.2012.11.022. Epub 2013 Jan 7. PMID 23305721
- [Background] Booya F, Bandarian F, Larijani B, Pajouhi M, Nooraei M, Lotfi J. Potential risk factors for diabetic neuropathy: a case control study. BMC Neurol. 2005 Dec 10;5:24. doi: 10.1186/1471-2377-5-24. PMID 16336693
- [Background] Borkosky SL, Roukis TS. Incidence of re-amputation following partial first ray amputation associated with diabetes mellitus and peripheral sensory neuropathy: a systematic review. Diabet Foot Ankle. 2012;3. doi: 10.3402/dfa.v3i0.12169. Epub 2012 Jan 20. PMID 22396832
- [Background] Casellini CM, Parson HK, Richardson MS, Nevoret ML, Vinik AI. Sudoscan, a noninvasive tool for detecting diabetic small fiber neuropathy and autonomic dysfunction. Diabetes Technol Ther. 2013 Nov;15(11):948-53. doi: 10.1089/dia.2013.0129. Epub 2013 Jul 27. PMID 23889506
- [Background] Chatterton BD, Muller S, Thomas MJ, Menz HB, Rome K, Roddy E. Inter and intra-rater repeatability of the scoring of foot pain drawings. J Foot Ankle Res. 2013 Nov 1;6(1):44. doi: 10.1186/1757-1146-6-44. PMID 24180324
- [Background] Chen L, Magliano DJ, Zimmet PZ. The worldwide epidemiology of type 2 diabetes mellitus--present and future perspectives. Nat Rev Endocrinol. 2011 Nov 8;8(4):228-36. doi: 10.1038/nrendo.2011.183. PMID 22064493
- [Background] Chyun DA, Melkus GD, Katten DM, Price WJ, Davey JA, Grey N, Heller G, Wackers FJ. The association of psychological factors, physical activity, neuropathy, and quality of life in type 2 diabetes. Biol Res Nurs. 2006 Apr;7(4):279-88. doi: 10.1177/1099800405285748. PMID 16581898
- [Background] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Background] Cox AA, Sagot Y, Hedou G, Grek C, Wilkes T, Vinik AI, Ghatnekar G. Low-Dose Pulsatile Interleukin-6 As a Treatment Option for Diabetic Peripheral Neuropathy. Front Endocrinol (Lausanne). 2017 May 2;8:89. doi: 10.3389/fendo.2017.00089. eCollection 2017. PMID 28512447
- [Background] Dixit S, Maiya A, Shastry B. Effect of aerobic exercise on quality of life in population with diabetic peripheral neuropathy in type 2 diabetes: a single blind, randomized controlled trial. Qual Life Res. 2014 Jun;23(5):1629-40. doi: 10.1007/s11136-013-0602-7. Epub 2013 Dec 11. PMID 24326731
- [Background] Fernando M, Crowther R, Lazzarini P, Sangla K, Cunningham M, Buttner P, Golledge J. Biomechanical characteristics of peripheral diabetic neuropathy: A systematic review and meta-analysis of findings from the gait cycle, muscle activity and dynamic barefoot plantar pressure. Clin Biomech (Bristol). 2013 Oct;28(8):831-45. doi: 10.1016/j.clinbiomech.2013.08.004. Epub 2013 Aug 27. PMID 24035444
- [Background] Ferreira JP, Sartor CD, Leal AM, Sacco IC, Sato TO, Ribeiro IL, Soares AS, Cunha JE, Salvini TF. The effect of peripheral neuropathy on lower limb muscle strength in diabetic individuals. Clin Biomech (Bristol). 2017 Mar;43:67-73. doi: 10.1016/j.clinbiomech.2017.02.003. Epub 2017 Feb 9. PMID 28213167
- [Background] Glatte P, Buchmann SJ, Hijazi MM, Illigens BM, Siepmann T. Architecture of the Cutaneous Autonomic Nervous System. Front Neurol. 2019 Sep 10;10:970. doi: 10.3389/fneur.2019.00970. eCollection 2019. PMID 31551921
- [Background] Holloszy JO. Exercise-induced increase in muscle insulin sensitivity. J Appl Physiol (1985). 2005 Jul;99(1):338-43. doi: 10.1152/japplphysiol.00123.2005. PMID 16036907
- [Background] Kelly C, Fleischer A, Yalla S, Grewal GS, Albright R, Berns D, Crews R, Najafi B. Fear of falling is prevalent in older adults with diabetes mellitus but is unrelated to level of neuropathy. J Am Podiatr Med Assoc. 2013 Nov-Dec;103(6):480-8. doi: 10.7547/1030480. PMID 24297984
- [Background] Kukidome D, Nishikawa T, Sato M, Nishi Y, Shimamura R, Kawashima J, Shimoda S, Mizuta H, Araki E. Impaired balance is related to the progression of diabetic complications in both young and older adults. J Diabetes Complications. 2017 Aug;31(8):1275-1282. doi: 10.1016/j.jdiacomp.2017.05.014. Epub 2017 Jun 4. PMID 28610947
- [Background] Leelarungrayub D, Saidee K, Pothongsunun P, Pratanaphon S, YanKai A, Bloomer RJ. Six weeks of aerobic dance exercise improves blood oxidative stress status and increases interleukin-2 in previously sedentary women. J Bodyw Mov Ther. 2011 Jul;15(3):355-62. doi: 10.1016/j.jbmt.2010.03.006. Epub 2010 Apr 28. PMID 21665113
- [Background] Morrison S, Colberg SR, Parson HK, Vinik AI. Exercise improves gait, reaction time and postural stability in older adults with type 2 diabetes and neuropathy. J Diabetes Complications. 2014 Sep-Oct;28(5):715-22. doi: 10.1016/j.jdiacomp.2014.04.007. Epub 2014 Apr 18. PMID 24929798
- [Background] Mueller MJ, Tuttle LJ, Lemaster JW, Strube MJ, McGill JB, Hastings MK, Sinacore DR. Weight-bearing versus nonweight-bearing exercise for persons with diabetes and peripheral neuropathy: a randomized controlled trial. Arch Phys Med Rehabil. 2013 May;94(5):829-38. doi: 10.1016/j.apmr.2012.12.015. Epub 2012 Dec 28. PMID 23276801
- [Background] Muller KA, Ryals JM, Feldman EL, Wright DE. Abnormal muscle spindle innervation and large-fiber neuropathy in diabetic mice. Diabetes. 2008 Jun;57(6):1693-701. doi: 10.2337/db08-0022. Epub 2008 Mar 24. PMID 18362211
- [Background] Noopud P, Suputtitada A, Khongprasert S, Kanungsukkasem V. Effects of Thai traditional dance on balance performance in daily life among older women. Aging Clin Exp Res. 2019 Jul;31(7):961-967. doi: 10.1007/s40520-018-1040-8. Epub 2018 Oct 8. PMID 30298380
- [Background] Oh TJ, Kang S, Lee JE, Moon JH, Choi SH, Lim S, Jang HC. Association between deterioration in muscle strength and peripheral neuropathy in people with diabetes. J Diabetes Complications. 2019 Aug;33(8):598-601. doi: 10.1016/j.jdiacomp.2019.04.007. Epub 2019 Apr 13. PMID 31129004
- [Background] Okada S, Hiuge A, Makino H, Nagumo A, Takaki H, Konishi H, Goto Y, Yoshimasa Y, Miyamoto Y. Effect of exercise intervention on endothelial function and incidence of cardiovascular disease in patients with type 2 diabetes. J Atheroscler Thromb. 2010 Aug 31;17(8):828-33. doi: 10.5551/jat.3798. Epub 2010 May 13. PMID 20467191
- [Background] Hewston P, Deshpande N. Fear of Falling and Balance Confidence in Older Adults With Type 2 Diabetes Mellitus: A Scoping Review. Can J Diabetes. 2018 Dec;42(6):664-670. doi: 10.1016/j.jcjd.2018.02.009. Epub 2018 Mar 6. PMID 29914779
- [Background] Pirker W, Katzenschlager R. Gait disorders in adults and the elderly : A clinical guide. Wien Klin Wochenschr. 2017 Feb;129(3-4):81-95. doi: 10.1007/s00508-016-1096-4. Epub 2016 Oct 21. PMID 27770207
- [Background] Plagemann A, Heidrich I, Gotz F, Rohde W, Dorner G. Obesity and enhanced diabetes and cardiovascular risk in adult rats due to early postnatal overfeeding. Exp Clin Endocrinol. 1992;99(3):154-8. doi: 10.1055/s-0029-1211159. PMID 1526266
- [Background] Pop-Busui R, Boulton AJ, Feldman EL, Bril V, Freeman R, Malik RA, Sosenko JM, Ziegler D. Diabetic Neuropathy: A Position Statement by the American Diabetes Association. Diabetes Care. 2017 Jan;40(1):136-154. doi: 10.2337/dc16-2042. No abstract available. PMID 27999003
- [Background] Raymond B, Steriovski J, Gillyard K, Yang C, Wu SC, Crews RT. Choosing a Vibratory Test to Pair With Semmes Weinstein Monofilament Testing for Evaluating Lower Extremity Sensation in Patients With Diabetes: A Comparison of Three Vibratory Methodologies. J Diabetes Sci Technol. 2020 Jan;14(1):8-15. doi: 10.1177/1932296819849478. Epub 2019 May 21. PMID 31113243
- [Background] Seferovic JP, Pfeffer MA, Claggett B, Desai AS, de Zeeuw D, Haffner SM, McMurray JJV, Parving HH, Solomon SD, Chaturvedi N. Three-question set from Michigan Neuropathy Screening Instrument adds independent prognostic information on cardiovascular outcomes: analysis of ALTITUDE trial. Diabetologia. 2018 Mar;61(3):581-588. doi: 10.1007/s00125-017-4485-y. Epub 2017 Nov 3. PMID 29098323
- [Background] Spink MJ, Fotoohabadi MR, Menz HB. Foot and ankle strength assessment using hand-held dynamometry: reliability and age-related differences. Gerontology. 2010;56(6):525-32. doi: 10.1159/000264655. Epub 2009 Dec 3. PMID 19955706
- [Background] Sun PC, Lin HD, Jao SH, Chan RC, Kao MJ, Cheng CK. Thermoregulatory sudomotor dysfunction and diabetic neuropathy develop in parallel in at-risk feet. Diabet Med. 2008 Apr;25(4):413-8. doi: 10.1111/j.1464-5491.2008.02395.x. Epub 2008 Mar 13. PMID 18341593
- [Background] Turner G, Quigg S, Davoren P, Basile R, McAuley SA, Coombes JS. Resources to Guide Exercise Specialists Managing Adults with Diabetes. Sports Med Open. 2019 Jun 3;5(1):20. doi: 10.1186/s40798-019-0192-1. PMID 31161377
- [Background] van Deursen RW, Simoneau GG. Foot and ankle sensory neuropathy, proprioception, and postural stability. J Orthop Sports Phys Ther. 1999 Dec;29(12):718-26. doi: 10.2519/jospt.1999.29.12.718. PMID 10612069
- [Background] van Praag H, Shubert T, Zhao C, Gage FH. Exercise enhances learning and hippocampal neurogenesis in aged mice. J Neurosci. 2005 Sep 21;25(38):8680-5. doi: 10.1523/JNEUROSCI.1731-05.2005. PMID 16177036